CLINICAL TRIAL: NCT03962751
Title: Motivating Campus Change (MC2) Project Pilot Study
Brief Title: Motivating Campus Change Project Pilot Study
Acronym: MC2 Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Mary Larimer, Professor, School of Medicine, Psychiatry and Behavioral Sciences, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00004630; R01AA012547-11A1 (NIH); R56AA012547-11A1 (NIH)
Record Dates: First submitted 2019-05-08; First posted 2019-05-24 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Drinking Behavior
MeSH Terms: conditions — Drinking Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Sequential Post Feedback Information Delivery (Experimental): Participants receive the first component of their PFI immediately following Baseline and subsequently receive 1 component each week until they receive all 4 components. Participants will complete a Post Feedback Survey and a 3 week follow back and Knowledge assessment.
  Interventions: Behavioral: Sequential Post Feedback Intervention Delivery
- Sequential Post Feedback Information Delivery +Text Messages (Experimental): Participants receive the first component of their PFI immediately following Baseline and subsequently receive 1 component each week until they receive all 4 components. Participants will complete a Post Feedback Survey and a 3 week follow back and Knowledge assessment. Additionally, participants receive the Text Message Booster Component in the days before and during their birthday celebration(s).
  Interventions: Behavioral: Sequential Post Feedback Intervention Delivery; Behavioral: Text Message Boosters
- Simultaneous Post Feedback Information Delivery (Experimental): Participants receive all 4 feedback components immediately after providing consent to the Pilot Feasibility Study following the Screening/Baseline Survey. Participants complete a brief 10 minute Post-Feedback Survey and a 3 Week Followup Survey to assess knowledge of the intervention feedback content.
  Interventions: Behavioral: Simultaneous Post Feedback Intervention Delivery
- Simultaneous Post Feedback Information Delivery +Text Messages (Experimental): Participants receive all 4 feedback components immediately after providing consent to the Pilot Feasibility Study following the Screening/Baseline Survey. Participants complete a brief 10 minute Post-Feedback Survey and a 3 Week Followup Survey to assess knowledge of the intervention feedback content. Additionally, participants receive the Text Message Booster Component in the days before and during their birthday celebration(s).
  Interventions: Behavioral: Simultaneous Post Feedback Intervention Delivery; Behavioral: Text Message Boosters
- Baseline Assessment Only (No Intervention): Participants complete baseline survey and conclude participation.

INTERVENTIONS:
Behavioral: Simultaneous Post Feedback Intervention Delivery — Simultaneous PFI delivery after baseline survey
  Arms: Simultaneous Post Feedback Information Delivery; Simultaneous Post Feedback Information Delivery +Text Messages
Behavioral: Sequential Post Feedback Intervention Delivery — Sequential PFI delivery over 3 weeks after baseline survey
  Arms: Sequential Post Feedback Information Delivery; Sequential Post Feedback Information Delivery +Text Messages
Behavioral: Text Message Boosters — Text message boosters on PFI content during week of high risk drinking event
  Arms: Sequential Post Feedback Information Delivery +Text Messages; Simultaneous Post Feedback Information Delivery +Text Messages

SUMMARY:
This study tests the optimization and delivery feasibility of personalized feedback interventions to address harmful alcohol use among college students.

DETAILED DESCRIPTION:
This study builds upon the latest alcohol intervention literature to develop and test the next wave of personalized feedback interventions (PFIs) to address harmful alcohol use among college students. The purpose of this research is to determine optimal configuration of PFIs to take advantage of the clarity and initial impact of single-component PFIs and greater effect size and duration of personalized multi-component PFIs. The Investigators seek to increase and evaluate engagement with the PFI and text-message materials and boost innovation of both content and process of the intervention. In addition to PFI content and delivery, the investigators will use qualitative and quantitative methods to determine personal relevance of the chosen high-risk events among a sample of students who engage in heavy episodic drinking to better understand duration of PFI effects impacted by fluctuations in drinking associated with high-risk events. Prior interventions have targeted drinking in general or a single high-risk drinking event (e.g., Spring Break), but have not targeted both general and event-specific drinking together. These enhanced intervention effects, could have a significant impact on risks associated with college student drinking, and can be rapidly disseminated and implemented on campuses nationwide to address the public health problem posed by heavy episodic drinking among college students.

This study conducts a screening/baseline assessment to collect quantitative data on high risk drinking situations and related norms and screens participants for eligibility for the Pilot Feasibility Study. The purpose of the Pilot Feasibility Study is to test the feasibility of sending participants web-based personalized feedback targeting their general drinking behavior in a single dose (Simultaneous) versus broken up into 4 components administered one week apart (Sequential) with half of participants in each group also being randomly selected to receive a text message booster component targeting drinking during their upcoming birthday celebration.

ELIGIBILITY:
Inclusion Criteria:

* birthday that falls withing summer/ fall 2018 assessment window
* at least 1 heavy episodic drinking episode in the past month
* at least 3 negative alcohol related consequences on Rutgers Alcohol Problem Index/ Young Adult Alcohol Problems Screening Test in the past 3 months
* intend to consume alcohol over the week of their birthday
* Indicate they own a cell phone with text message capabilities and consent to receiving text messages

Exclusion Criteria:

* Doesn't meet inclusion criteria
* Unwillingness to participate
* Failure to provide consent

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 250 (Actual)
Dates: Start 2018-06-28 (Actual); Primary Completion 2018-11-04 (Actual); Study Completion 2018-11-04 (Actual)

PRIMARY OUTCOMES:
Satisfaction with different modes of delivery of personalized information on health behaviors | 2-3 months of intervention assessment
  The primary outcome of this program of research is to assess participant satisfaction of different modes of personalized information delivery. The participants receive personalized information related to health behaviors all at once or weekly over the course of 4 weeks and satisfaction is assessed using survey completion rates, tracked interaction with the personalized feedback information, and a series of satisfaction related questions.

CONTACTS AND LOCATIONS:
Overall Officials: Mary E Larimer, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States